CLINICAL TRIAL: NCT04699045
Title: Prenatal Iron Status and Its Association With Cord Blood and Infant Ferritin Level
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: Ferritin_cohort
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No active intervention

SUMMARY:
Iron deficiency (ID) in early life is associated with significant morbidities. Most fetal iron required for infant growth is acquired in the third trimester from maternal iron store. However, how prenatal iron level affects newborn's ferritin level at birth and in early infancy remains controversial. This study aimed to examine the associations between maternal ferritin levels with cord blood serum ferritin (CBSF) and to compare the ferritin levels between different feeding practices in early infancy.

DETAILED DESCRIPTION:
Iron deficiency (ID) is the most common micronutrient deficiency globally. Pregnant women and young children are at risk of ID. During pregnancy, there is an increased demand for iron to accommodate the needs of the fetal-placental unit. This increase in physiologic demand for iron renders pregnant women vulnerable to ID. In fact, ID is the major cause of anemia in pregnancy and can increase the perinatal maternal morbidity and mortality. Iron is also an essential micronutrient for fetal and infant brain development. ID in early life is associated with worse cognitive, motor, social emotional as well as neurophysiological development. Besides neurodevelopment, iron is also essential for proper immune function affecting both innate and adaptive cell, and has implications for childhood atopic diseases.

Globally, there is an increasing trend of breastfeeding especially in developed countries.In Hong Kong, the government's continuing effort to promote breastfeeding has successfully boosted the rate of babies being breastfed. This encouraging information means more children will benefit from the many advantages of breast milk over formula milk, yet exclusive breastfeeding, particularly in the context of maternal ID and late weaning, may be a risk factor of ID in the infants. In view of the adverse impact of fetal and infant ID on neurocognitive development, it is important to evaluate the iron status of young infants, the effect of feeding practices on development of ID and the risk factors of ID in early infancy.

Maternal ID is prevalent worldwide varying from 20% to 90%. Previous investigation performed in the Department of Obstetrics and Gynaecology, Prince of Wales Hospital, concurred a significant prevalence (39%) of ID (serum ferritin < 15 microgram/L) among 100 asymptomatic pregnant women. Most fetal iron needed for infant growth is acquired in the third trimester from maternal iron store, in preparation for the high growth rate in the first 6 months of life. Iron status at birth is therefore critical and impaired iron status may persist into early childhood. However, low maternal prenatal iron levels measured as serum ferritin have not been consistently linked with low cord blood serum ferritin (CBSF) concentrations. Some studies reported that there was no correlation between serum ferritin of mothers and babies. However, others found that maternal ID or anemia, especially the severe type, adversely affected cord blood or infant iron status. Further studies are needed to evaluate how prenatal maternal iron status affects newborn's ferritin level at birth. Such data is necessary to guide future recommendations regarding the need of iron supplement in pregnant or lactating women and/or their infants. Hence, this study aimed to examine the associations between maternal prenatal ferritin levels with CBSF and to compare the ferritin levels with different feeding practices in early infancy at 3 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Women who carried a singleton pregnancy without any history of thyroid dysfunction, hyperemesis gravidarum, autoimmune disease, or any other major medical condition with cord blood available were eligible for this study

Exclusion Criteria:

* multiple pregnancy, preterm delivery at less than 37 weeks of gestation, infants with congenital anomalies, syndromal diseases, chronic renal or hepatic diseases, metabolic disease, chronic gastrointestinal diseases and/or malabsorption

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Chinese mothers with uncomplicated pregnancy were recruited from a cohort which was established to evaluate gestational age specific thyroid function during pregnancy. Between July 2014 and January 2016, pregnant women attended antenatal care in their first trimester of pregnancy were recruited by research personnel in the antenatal clinic at the Prince of Wales Hospital, which is a tertiary teaching hospital in Hong Kong. After delivery, mothers were again approached and invited to join this study by research personnel in the postnatal ward.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Ferritin concentrations | up to 3 months
  Ferritin concentrations in late pregnancy, in cord blood and in early infancy

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No